CLINICAL TRIAL: NCT07156058
Title: MiniPDX-based Postoperative Adjuvant Therapy for Biliary Tract Cancer: A Prospective Cohort Study
Brief Title: MiniPDX-based Postoperative Adjuvant Therapy for Biliary Tract Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2022A04
Record Dates: First submitted 2023-09-13; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MiniPDX group (Experimental): 102 patients with BTC after surgery will be treated with drugs or regimens tested by MiniPDX assays.
  Interventions: Other: MiniPDX group
- Treatment of Physician's Choice (TPC) (Active Comparator): TPC will be administered per standard of care. 102 patients after surgery in the same period will receive chemotherapy.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Other: MiniPDX group — Personalized treatment for guided by mini-PDX. The MiniPDX test can provide drug sensitivity results in as little as 7 days. Drugs including but not limited to the following agents: capecitabine, gemcitabine + cis-platinum, gemcitabine + capecitabine, 5-FU + oxaliplatin, gemcitabine, 5-FU, capecitabine + cis-platinum, 5-FU + cis-platinum.
  Arms: MiniPDX group
Drug: Capecitabine — Drug: Capecitabine
  Arms: Treatment of Physician's Choice (TPC)

SUMMARY:
This research aims to study the effect of postoperative adjuvant therapy with a MiniPDX drug sensitivity test for biliary tract cancer.

DETAILED DESCRIPTION:
Biliary tract cancer (BTC) is the most common primary malignancy of the biliary tract. Currently, surgery provides the only ray of hope for the management of BTC, however, the disease is progressing rapidly, lacking of obvious symptoms in its early stages, with metastases to lymph nodes. Only 20-30% of patients are eligible for surgical resection with curative intent. In addition, the treatment remains difficult because of the lack of effective chemotherapeutic agents and the combined regimens for reference.

In this study, fresh tumor samples generated directly from patients will be used for a MiniPDX test and inoculated in mice subcutaneously. The candidate drugs or regimens can be tested in mice to determine the best treatment for that specific patient after surgery.

The study aims to evaluate the efficacy and accuracy of MiniPDX assays for antitumor chemotherapeutics.

ELIGIBILITY:
Inclusion Criteria:

1. histologically documented biliary duct cancer (including intrahepatic cholangiocarcinoma, hilar cholangiocarcinoma, distal cholangiocarcinoma and gallbladder carcinoma). Patients underwent R0 resection.
2. Ambulatory male or female. Age ≥ 18 years.
3. ECOG performance status between 0 and 2
4. Patients must be tolerated with combination treatment with life expectancy of greater than 6 months.
5. No dysfunction and bleeding tendency in main organs (heart, liver, brain and kidneys); No history of blood disease; No cardiac insufficiency or chest pain (medically uncontrollable). No myocardial infarction occurred within 12 months before the start of the study.
6. Subjects must have normal organ as defined below: Hb ≥80 g/L; ANC ≥1.5×109/L; Platelets ≥100×109/L; AL/AST ≤2.5 x institutional upper limit of normal; ALP ≤2.5 x ULN; Total bilirubin <1.5 x ULN; Creatinine <1 x ULN; Serum albumin ≥30g/L.
7. Women of child-bearing potential must agree to use adequate contraception (IUD, contraceptives or condoms) for the duration of study participation, and for 6 months after completion of study; Serum or urine pregnancy tests are negative within 7 days before study entry; men must agree to use adequate contraception for the duration of study participation, and for 6 months after completion of study.
8. Patients must be willing to and able to follow the protocol during study entry.
9. Patients must be willing to sign an informed consent and able to understand that anytime is all right to quit the study without loss.

Exclusion Criteria:

1. Prior chemotherapy or radiotherapy.
2. Patients are in other clinical trials.
3. Coagulation disorders, history of blood disease or serious (active) heart disease such as coronary heart disease with apparent symptom, congestive heart failure of NYHA Class II or more severe, serious heart rhythm controlled by medicaments, or the attack of myocardial infarction within 12 months.
4. Hepatic and renal insufficiency with apparent symptom.
5. Pregnant or lactating female, or women of child-bearing age who have a positive serum pregnancy test or no tests. Female subjects of non-reproductive potential with post-menopausal for ≥1 year.
6. Patients with multiple primary cancer, or brain or meningeal metastases.
7. Patients with a history of uncontrolled epilepsy, central nervous system disease or mental disorder whose clinical severity, as judged by the investigator, may hinder the signing of informed consent or affect the patient's compliance with oral medication
8. Patients who need immunotherapy for organ transplantation.
9. Patients with recurrent infections, or other uncontrolled accompanying diseases, or hepatic cirrhosis caused hepatic injury or chronic active hepatitis (ALT ≥2 ULN, AST ≥1.5 ULN, PT >13 S or TB ≥2 ULN)
10. Moderate or severe kidney injury [CrCl ≤50 ml/min (Cockcroft-Gault Equation)], or creatinine > ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival (RFS) | Through study completion, an expected average of 2 year.
  The interval from surgery to diagnosis of recurrence in the patients enrolled.

SECONDARY OUTCOMES:
Overall Survival (OS) | Through study completion, an expected average of 2 year.
  The interval from randomization until death, whichever comes first.
Event-Free Survival (EFS) | Through study completion, an expected average of 2 year.
  The time from randomization to initial occurrence (including local recurrence, metastasis, second primary cancer, death or any cause among the above), whichever comes first.
Non-recurrence after radical surgery for BTC in 2 years | Through study completion, an expected average of 2 year.
  The ratio of patients with BTC after radical surgery without recurrence in 2 years.
Quality of Life (QOL) | Through study completion, an expected average of 2 year.
  Assessed by the EORTC QLQ-C30 for patients over 16 years old) or the Pediatric Quality of Life Inventory (PedsQL) for patients under 16 years old.

CONTACTS AND LOCATIONS:
Overall Officials: Xinyu Bi, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Background] Valle JW, Kelley RK, Nervi B, Oh DY, Zhu AX. Biliary tract cancer. Lancet. 2021 Jan 30;397(10272):428-444. doi: 10.1016/S0140-6736(21)00153-7. PMID 33516341
- [Background] Mizrahi JD, Shroff RT. New Treatment Options for Advanced Biliary Tract Cancer. Curr Treat Options Oncol. 2020 Jun 29;21(8):63. doi: 10.1007/s11864-020-00767-3. PMID 32602010
- [Background] Mondaca S, Nervi B, Pinto M, Abou-Alfa GK. Biliary tract cancer prognostic and predictive genomics. Chin Clin Oncol. 2019 Aug;8(4):42. doi: 10.21037/cco.2019.07.06. Epub 2019 Jul 29. PMID 31431036
- [Background] Nara S, Esaki M, Ban D, Takamoto T, Shimada K, Ioka T, Okusaka T, Ishii H, Furuse J. Adjuvant and neoadjuvant therapy for biliary tract cancer: a review of clinical trials. Jpn J Clin Oncol. 2020 Dec 16;50(12):1353-1363. doi: 10.1093/jjco/hyaa170. PMID 33037430
- [Background] Bridgewater JA, Goodman KA, Kalyan A, Mulcahy MF. Biliary Tract Cancer: Epidemiology, Radiotherapy, and Molecular Profiling. Am Soc Clin Oncol Educ Book. 2016;35:e194-203. doi: 10.1200/EDBK_160831. PMID 27249723
- [Background] Persano M, Puzzoni M, Ziranu P, Pusceddu V, Lai E, Pretta A, Donisi C, Pinna G, Spanu D, Cimbro E, Parrino A, Liscia N, Mariani S, Dubois M, Migliari M, Scartozzi M. Molecular-driven treatment for biliary tract cancer: the promising turning point. Expert Rev Anticancer Ther. 2021 Nov;21(11):1253-1264. doi: 10.1080/14737140.2021.1982699. Epub 2021 Sep 24. PMID 34551663
- [Background] Lamarca A, Barriuso J, McNamara MG, Valle JW. Molecular targeted therapies: Ready for "prime time" in biliary tract cancer. J Hepatol. 2020 Jul;73(1):170-185. doi: 10.1016/j.jhep.2020.03.007. Epub 2020 Mar 12. PMID 32171892
- [Background] Scott AJ, Sharman R, Shroff RT. Precision Medicine in Biliary Tract Cancer. J Clin Oncol. 2022 Aug 20;40(24):2716-2734. doi: 10.1200/JCO.21.02576. Epub 2022 Jul 15. PMID 35839428
- [Background] Zhang F, Wang W, Long Y, Liu H, Cheng J, Guo L, Li R, Meng C, Yu S, Zhao Q, Lu S, Wang L, Wang H, Wen D. Characterization of drug responses of mini patient-derived xenografts in mice for predicting cancer patient clinical therapeutic response. Cancer Commun (Lond). 2018 Sep 26;38(1):60. doi: 10.1186/s40880-018-0329-5. PMID 30257718
- [Background] Raja FA, Counsell N, Colombo N, Pfisterer J, du Bois A, Parmar MK, Vergote IB, Gonzalez-Martin A, Alberts DS, Plante M, Torri V, Ledermann JA. Platinum versus platinum-combination chemotherapy in platinum-sensitive recurrent ovarian cancer: a meta-analysis using individual patient data. Ann Oncol. 2013 Dec;24(12):3028-34. doi: 10.1093/annonc/mdt406. Epub 2013 Nov 4. PMID 24190964
- [Background] Vlachogiannis G, Hedayat S, Vatsiou A, Jamin Y, Fernandez-Mateos J, Khan K, Lampis A, Eason K, Huntingford I, Burke R, Rata M, Koh DM, Tunariu N, Collins D, Hulkki-Wilson S, Ragulan C, Spiteri I, Moorcraft SY, Chau I, Rao S, Watkins D, Fotiadis N, Bali M, Darvish-Damavandi M, Lote H, Eltahir Z, Smyth EC, Begum R, Clarke PA, Hahne JC, Dowsett M, de Bono J, Workman P, Sadanandam A, Fassan M, Sansom OJ, Eccles S, Starling N, Braconi C, Sottoriva A, Robinson SP, Cunningham D, Valeri N. Patient-derived organoids model treatment response of metastatic gastrointestinal cancers. Science. 2018 Feb 23;359(6378):920-926. doi: 10.1126/science.aao2774. PMID 29472484
- [Background] Lee SH, Hu W, Matulay JT, Silva MV, Owczarek TB, Kim K, Chua CW, Barlow LJ, Kandoth C, Williams AB, Bergren SK, Pietzak EJ, Anderson CB, Benson MC, Coleman JA, Taylor BS, Abate-Shen C, McKiernan JM, Al-Ahmadie H, Solit DB, Shen MM. Tumor Evolution and Drug Response in Patient-Derived Organoid Models of Bladder Cancer. Cell. 2018 Apr 5;173(2):515-528.e17. doi: 10.1016/j.cell.2018.03.017. PMID 29625057
- [Background] Sachs N, de Ligt J, Kopper O, Gogola E, Bounova G, Weeber F, Balgobind AV, Wind K, Gracanin A, Begthel H, Korving J, van Boxtel R, Duarte AA, Lelieveld D, van Hoeck A, Ernst RF, Blokzijl F, Nijman IJ, Hoogstraat M, van de Ven M, Egan DA, Zinzalla V, Moll J, Boj SF, Voest EE, Wessels L, van Diest PJ, Rottenberg S, Vries RGJ, Cuppen E, Clevers H. A Living Biobank of Breast Cancer Organoids Captures Disease Heterogeneity. Cell. 2018 Jan 11;172(1-2):373-386.e10. doi: 10.1016/j.cell.2017.11.010. Epub 2017 Dec 7. PMID 29224780
- [Background] Bruna A, Rueda OM, Greenwood W, Batra AS, Callari M, Batra RN, Pogrebniak K, Sandoval J, Cassidy JW, Tufegdzic-Vidakovic A, Sammut SJ, Jones L, Provenzano E, Baird R, Eirew P, Hadfield J, Eldridge M, McLaren-Douglas A, Barthorpe A, Lightfoot H, O'Connor MJ, Gray J, Cortes J, Baselga J, Marangoni E, Welm AL, Aparicio S, Serra V, Garnett MJ, Caldas C. A Biobank of Breast Cancer Explants with Preserved Intra-tumor Heterogeneity to Screen Anticancer Compounds. Cell. 2016 Sep 22;167(1):260-274.e22. doi: 10.1016/j.cell.2016.08.041. Epub 2016 Sep 15. PMID 27641504
- [Background] Marangoni E, Vincent-Salomon A, Auger N, Degeorges A, Assayag F, de Cremoux P, de Plater L, Guyader C, De Pinieux G, Judde JG, Rebucci M, Tran-Perennou C, Sastre-Garau X, Sigal-Zafrani B, Delattre O, Dieras V, Poupon MF. A new model of patient tumor-derived breast cancer xenografts for preclinical assays. Clin Cancer Res. 2007 Jul 1;13(13):3989-98. doi: 10.1158/1078-0432.CCR-07-0078. PMID 17606733
- [Background] Friedman AA, Letai A, Fisher DE, Flaherty KT. Precision medicine for cancer with next-generation functional diagnostics. Nat Rev Cancer. 2015 Dec;15(12):747-56. doi: 10.1038/nrc4015. Epub 2015 Nov 5. PMID 26536825
- [Background] Ricci F, Bizzaro F, Cesca M, Guffanti F, Ganzinelli M, Decio A, Ghilardi C, Perego P, Fruscio R, Buda A, Milani R, Ostano P, Chiorino G, Bani MR, Damia G, Giavazzi R. Patient-derived ovarian tumor xenografts recapitulate human clinicopathology and genetic alterations. Cancer Res. 2014 Dec 1;74(23):6980-90. doi: 10.1158/0008-5472.CAN-14-0274. Epub 2014 Oct 10. PMID 25304260
- [Background] Zhan M, Yang RM, Wang H, He M, Chen W, Xu SW, Yang LH, Liu Q, Long MM, Wang J. Guided chemotherapy based on patient-derived mini-xenograft models improves survival of gallbladder carcinoma patients. Cancer Commun (Lond). 2018 Jul 17;38(1):48. doi: 10.1186/s40880-018-0318-8. PMID 30016995
- [Background] Solaini L, Jamieson NB, Metcalfe M, Abu Hilal M, Soonawalla Z, Davidson BR, McKay C, Kocher HM; UK Duodenal Cancer Study Group. Outcome after surgical resection for duodenal adenocarcinoma in the UK. Br J Surg. 2015 May;102(6):676-81. doi: 10.1002/bjs.9791. Epub 2015 Mar 16. PMID 25776995
- [Background] Zhao P, Chen H, Wen D, Mou S, Zhang F, Zheng S. Personalized treatment based on mini patient-derived xenografts and WES/RNA sequencing in a patient with metastatic duodenal adenocarcinoma. Cancer Commun (Lond). 2018 Aug 23;38(1):54. doi: 10.1186/s40880-018-0323-y. PMID 30139386
- [Background] Yang L, Yuan Z, Zhang Y, Cui Z, Li Y, Hou J, Liu X, Liu Z, Shi R, Tian Q, Wang J, Wang L. MiniPDX-guided postoperative anticancer treatment can effectively prolong the survival of patients with hepatocellular carcinoma. Cancer Chemother Pharmacol. 2021 Jan;87(1):125-134. doi: 10.1007/s00280-020-04182-1. Epub 2020 Nov 3. PMID 33141330
- [Background] Huang Y, Xu J, Li K, Wang J, Dai Y, Kang Y. A Novel, Personalized Drug-Screening System for Platinum-Resistant Ovarian Cancer Patients: A Preliminary Clinical Report. Cancer Manag Res. 2021 Mar 29;13:2849-2867. doi: 10.2147/CMAR.S276799. eCollection 2021. PMID 33833569
- [Background] Li C, Sun YD, Yu GY, Cui JR, Lou Z, Zhang H, Huang Y, Bai CG, Deng LL, Liu P, Zheng K, Wang YH, Wang QQ, Li QR, Wu QQ, Liu Q, Shyr Y, Li YX, Chen LN, Wu JR, Zhang W, Zeng R. Integrated Omics of Metastatic Colorectal Cancer. Cancer Cell. 2020 Nov 9;38(5):734-747.e9. doi: 10.1016/j.ccell.2020.08.002. Epub 2020 Sep 3. PMID 32888432
- [Background] Wang J, Sun T, Meng Z, Wang L, Li M, Chen J, Qin T, Yu J, Zhang M, Bie Z, Dong Z, Jiang X, Lin L, Zhang C, Liu Z, Jiang R, Yang G, Li L, Zhang Y, Huang D. XPO1 inhibition synergizes with PARP1 inhibition in small cell lung cancer by targeting nuclear transport of FOXO3a. Cancer Lett. 2021 Apr 10;503:197-212. doi: 10.1016/j.canlet.2021.01.008. Epub 2021 Jan 23. PMID 33493586
- [Background] Wang X, Sun Y, Xu Y, Wen D, An N, Leng X, Fu G, Lu S, Chen Z. Mini-patient-derived xenograft assay based on microfluidic technology promises to be an effective tool for screening individualized chemotherapy regimens for advanced non-small cell lung cancer. Cell Biol Int. 2021 Sep;45(9):1887-1896. doi: 10.1002/cbin.11622. Epub 2021 Jun 26. PMID 33945662